CLINICAL TRIAL: NCT00122408
Title: Effect of Enterally Administered Probiotics in Mechanically Ventilated Patients: Double-Blind, Prospective Randomized Study Versus Placebo
Brief Title: Probiotic Enteral Administration in Mechanically Ventilated Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Mr P Boulanger / Directeur de la Recherche et de l'innovation, CHU Nancy
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: promotion_070605-gibot_DRI
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Pneumonia
Keywords: ventilator-associated pneumonia; probiotic; mechanical ventilation; intensive care
MeSH Terms: conditions — Pneumonia; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator)
  Interventions: Dietary Supplement: Ergyphilus
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: Ergyphilus

INTERVENTIONS:
Dietary Supplement: Ergyphilus — 5 pills a day of Ergyphilus or placebo

SUMMARY:
The objective of this study is to assess the effects of a daily enteral supplementation with probiotics within a population of critically ill, mechanically ventilated patients. Especially, the effects of probiotics on mortality rate in intensive care medicine will be analysed.

DETAILED DESCRIPTION:
In a critically ill patient, the gut integrity is rapidly compromised either by the treatments used (such as catecholamine or antibiotics) or by the disease itself. This gut alteration favours the adhesion and/or internalisation of bacteria by intestine cells which lead to the production of large amounts of cytokines that rapidly reach the blood compartment, inducing neutrophils activation and then organ damage. Moreover, the imbalance in the normal intestinal flora (demonstrated as early as 24 hours after ICU admission) is one of the mechanisms involved in the development of ventilator associated pneumonia (VAP). VAP is the leading cause of ICU-acquired infection and is responsible for prolonged ICU stay, increased mortality and costs. Probiotics, and especially Lactobacillus Rhamnosus GG ('LGG'), have been demonstrated to possess beneficial effects in terms of intestine flora imbalance and immune response.

Objective: To study the effects of a probiotic mixture (containing LGG) enteral administration on the survival and the incidence of VAP in mechanically ventilated patients.

Patients and Methods: Prospective, randomized, double-blind, placebo-controlled study. After randomization, 740 intubated patients with a predictive length of mechanical support of more than 48 hours will enterally receive either 10.10 cfu of probiotic (Ergyphilus, Nutergia, France) or a identical placebo daily until withdrawal of mechanical support. The main endpoint is the mortality rate in ICU. Secondary endpoints include hospital length of stay and mortality rate, VAP incidence and the number of days free from antibiotics. Length of the study 24 months.

Perspectives: The objective is to demonstrate a survival advantage due to LGG administration, along with a reduction of VAP episodes and antibiotic use.

ELIGIBILITY:
Inclusion Criteria:

* Patients under mechanical ventilation for at least 48 hours

Exclusion Criteria:

* Age under 18
* Pregnancy
* Immunocompromised status
* Short bowel disease
* Moribund condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740 (Estimated)
Dates: Start 2006-01; Primary Completion 2009-08 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Intensive Care Unit (ICU) mortality rate | 28 days

SECONDARY OUTCOMES:
Hospital mortality rate | 60 days
incidence of ventilator-associated pneumonia | 28 days
incidence of multi-resistant bacteria infection and colonization | 28 days
incidence of diarrhea | 28 days
ICU length of stay | 60 days
hospital length of stay | 60 days
antibiotic use in ICU (antibiotic-free days) | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Gibot, MD, PhD, Principal Investigator — CHU NANCY
Locations (3):
- France (3):
  - CHG, Mâcon
  - CHR, Metz
  - Hopital Central, Service de Reanimation Medicale, Nancy